CLINICAL TRIAL: NCT03832478
Title: Longitudinal Virtual Reality Use in Pediatric Surgical Procedures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical difficulty with sending device home with patients
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Stephanie D. Chao, Assistant Professor of Surgery (Pediatric Surgery), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 46879
Record Dates: First submitted 2019-01-23; First posted 2019-02-06 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Anxiety; Pain; Pain, Postoperative
Keywords: Virtual Reality; Meditation; Mindfulness Meditation; Guided Mindfulness Meditation; Anxiety; Pain; Postoperative pain
MeSH Terms: conditions — Anxiety Disorders; Pain; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Prospective observational study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Headset Given (Experimental): Virtual Reality headset (Samsung Gear VR) with mindfulness meditation app is given for patient use prior to surgery date and for duration of postoperative stay.
  Interventions: Device: Virtual Reality Headset Given

INTERVENTIONS:
Device: Virtual Reality Headset Given — Samsung Gear VR Headset with guided mindfulness meditation app

SUMMARY:
This study aims to investigate the use of virtual reality guided mindfulness meditation to reduce the pre and post-operative anxiety and pain of pediatric surgical patients.

DETAILED DESCRIPTION:
Pre-procedural anxiety in pediatric patients has been previously shown to increase the likelihood of family stressors, agitation, sleep disturbances, and negative behavioral changes. Post-procedural pain has been shown to negatively impact future interactions with healthcare personnel. The purpose of this study is to determine the feasibility of using guided mindfulness meditation through a non-invasive device (virtual reality headset) to manage pre-procedure anxiety and post-procedure anxiety and pain.

ELIGIBILITY:
Inclusion Criteria:

* Have parental consent if under 18 or 18 and older but unable to provide own consent
* Can comprehend instructions in English language
* Is undergoing surgical procedure requiring general anesthesia at Lucile Packard Children's Hospital
* Children that are normally healthy (ASA I) or have a mild systemic disease (ASA II, III)

Exclusion Criteria:

* Children with significant cognitive impairment or developmental delays per parental report or H&P
* Children with ASA IV (severe systemic disease that is a constant threat to life) or ASA V (unstable patients not expected to survive >24hours or without operation)
* Children currently taking psychotropic mediations will be excluded from this study due to the affect emotion modulation
* Children with history of seizures related to photosensitivity.

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Children's Fear Scale | Before and after every use of the app (from date of enrollment to surgical procedure, up to 8 weeks. If patient has not undergone surgical procedure by 8 weeks, participation in study will be concluded and subject censored during data analysis)
  The Children's Fear Scale (McMurty et al., 2011) is a self-report scale that uses cartoon depictions of faces to quantify on a 0-4 scale how scared a child is at the given moment.
Change in Faces Pain Scale | Before and after every use of the app (from date of enrollment to surgical procedure, up to 8 weeks. If patient has not undergone surgical procedure by 8 weeks, participation in study will be concluded and subject censored during data analysis)
  The Faces Pain Scale (Hicks et al., 2001) is a self-report scale that uses cartoon depictions of faces to quantify on a 0-10 scale how much pain a child is experiencing at the given moment.
Change in Anxiety Scale | Before and after every use of the app (from date of enrollment to surgical procedure, up to 8 weeks. If patient has not undergone surgical procedure by 8 weeks, participation in study will be concluded and subject censored during data analysis)
  A self-report question on a 1-5 scale will be asked to assess how much anxiety a child is experiencing at the given moment.

SECONDARY OUTCOMES:
Patient and Parent Satisfaction Surveys | Satisfaction surveys will be administered at the time of study completion (when the patient has completed his/her surgical procedure and is ready for hospital discharge/or 30 days post-procedure, whichever occurs first)
  Parents, and patients will be given self-report survey questions asking about their satisfaction with the technology, the patients' immersion with the technology, and desire for use in future procedures. Questions will be answered on a 1-5 scale .
Clinician Satisfaction Surveys | Satisfaction survey will be administered to physicians within 48 hours of procedure completion. Physicians may return surveys up to one month post-procedure.
  Surgeons and anesthesiologists will be given self-report survey questions asking about their satisfaction with the technology, the patients' immersion with the technology, and desire for use in future procedures. Questions will be answered on a 1-5 scale .

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie D Chao, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Stanford Pediatric Surgery Clinic, Palo Alto, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li A, Montano Z, Chen VJ, Gold JI. Virtual reality and pain management: current trends and future directions. Pain Manag. 2011 Mar;1(2):147-157. doi: 10.2217/pmt.10.15. PMID 21779307
- [Background] Won AS, Bailey J, Bailenson J, Tataru C, Yoon IA, Golianu B. Immersive Virtual Reality for Pediatric Pain. Children (Basel). 2017 Jun 23;4(7):52. doi: 10.3390/children4070052. PMID 28644422
- [Background] Zeidan F, Gordon NS, Merchant J, Goolkasian P. The effects of brief mindfulness meditation training on experimentally induced pain. J Pain. 2010 Mar;11(3):199-209. doi: 10.1016/j.jpain.2009.07.015. Epub 2009 Oct 22. PMID 19853530
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] He HG, Zhu L, Chan SW, Liam JL, Li HC, Ko SS, Klainin-Yobas P, Wang W. Therapeutic play intervention on children's perioperative anxiety, negative emotional manifestation and postoperative pain: a randomized controlled trial. J Adv Nurs. 2015 May;71(5):1032-43. doi: 10.1111/jan.12608. Epub 2015 Jan 6. PMID 25561079